CLINICAL TRIAL: NCT03897101
Title: Autophagy, Mitophagy, Inflammation and Plasmatic Concentration of Melatonin in Newborn With Metabolic Acidosis at Birth
Brief Title: Inflammation and Metabolic Acidosis at Birth (AGAIN: AutophaGy AcIdosis Newborn)
Acronym: AGAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Collaborators: AUSL Romagna Rimini (Other)
Responsible Party: Principal Investigator, Anna Tarocco, Medical Doctor, Principal Investigator, University Hospital of Ferrara
Other Study IDs: 639/2018/Sper/AOUFe
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Neonatal Encephalopathy; Cell Damage; Metabolic Acidosis; Inflammation
Keywords: mild neonatal encephalopathy; birth asphyxia; metabolic acidosis; Autophagy; Mitophagy; inflammation
MeSH Terms: conditions — Acidosis; Inflammation; Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MILD NE: gestational age > 35 weeks and weight > 1800 gr
  * Apgar score < 5 at 10 minutes o need for cardiopulmonary resuscitation at 10 minutes or evidence of base excess > 12 mmol/L or pH < 7,0 at initial blood gas analyses
  * evidence of mild encephalopathy graded according to Sarnat&Sarnat neurological evaluation
  * normal amplitude integrated electroencephalography
  Plasma levels of melatonin, Atg5, Parkin, Pink1, inflammatory cytokines will be evaluated
- ISOLATED METABOLIC ACIDOSIS: gestational age > 35 weeks and weight > 1800 gr
  * evidence of base excess > 12 mmol/L or pH < 7,0 at initial blood gas analyses
  * Normal Sarnat&Sarnat neurological evaluation
  Plasma levels of melatonin, Atg5, Parkin, Pink1, inflammatory cytokines will be evaluated
- HEALTY CONTROLS: gestational age > 35 weeks and weight > 1800 gr Normal blood pH or base excess
  Plasma levels of melatonin, Atg5, Parkin, Pink1, inflammatory cytokiness will be evaluated

SUMMARY:
Protection of brain development is a major aim in the Neonatal Intensive Care Unit. Neonatal encephalopathy (NE) occurs in 1.8 to 7.7 infants per 1000 births. Over the last six years, several randomized control trials have demonstrated that therapeutic hypothermia reduces the rate of death or disability at 18 months of age among infants who survived. However, the neurodevelopmental outcome in milder NE not treated with hypothermia remains unclear.

A multicenter prospective observational study will be conducted to determine biological changes of mild neonatal encephalopathy who are not recruited for therapeutic hypothermia .

DETAILED DESCRIPTION:
It is a prospective observational multicenter study on 50 newborns with mild neonatal encephalopathy and metabolic acidosis at birth not qualified for therapeutic hypothermia compared to healthy controls.

Infants with metabolic acidosis at birth and evidence of mild encephalopathy graded according to Sarnat&Sarnat neurological evaluation will be recruited to evaluate plasma concentration of melatonin and levels of Autophagy, mitophagy and inflammation.

Plasmatic changes will be compared to:

* healthy control
* infants with isolated metabolic acidosis at birth and normal neurological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* gestational age > 35 weeks and weight > 1800 gr
* Apgar score < 5 at 10 minutes o need for cardiopulmonary resuscitation at 10 minutes or evidence of base excess > 12 mmol/L or pH < 7,0 at initial blood gas analyses
* evidence of mild encephalopathy graded according to Sarnat&Sarnat neurological evaluation
* normal amplitude integrated electroencephalography

Exclusion Criteria:

* suspected inborn errors of metabolism
* major chromosomal congenital defects

Ages: 15 Minutes to 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: will be recruited 50 newborns with mild neonatal encephalopathy and metabolic acidosis at birth not qualified for therapeutic hypothermia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline ATG5 Plasma concentration at 7 days of life | birth, 72 hours, 7 days of life
  correlation between metabolic acidosis at birth and Autophagy. ELISA test will be used to measure plasma levels of ATG5

SECONDARY OUTCOMES:
change from baseline Parkin and Pink1 Plasma concentration at 7 days of life | birth, 72 hours, 7 days of life
  correlation between metabolic acidosis at birth and Mitophagy. ELISA test will be used to measure plasma levels of Parkin and Park1

OTHER OUTCOMES:
change from baseline Plasma Concentration of Melatonin at 7 days of life | birth, 72 hours, 7 days of life
  UPLC-Massa Acquity-Xevo TQD (Waters) will be used to measure plasma melatonin concentration.
change from baseline of inflammatory cytokines at 7 days of life | birth, 72 hours, 7 days of life
  correlation between metabolic acidosis at birth and inflammatory cytokines. ELISA test will be used to measure plasma levels inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Tarocco, MD, Principal Investigator — University Hospital s. Anna Ferrara
Locations (2):
- Italy (2):
  - University Hospital "Sant'Anna" of Ferrara, Ferrara
  - Infermi Hospital Rimini, Rimini

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alirezaei M, Kemball CC, Whitton JL. Autophagy, inflammation and neurodegenerative disease. Eur J Neurosci. 2011 Jan;33(2):197-204. doi: 10.1111/j.1460-9568.2010.07500.x. Epub 2010 Dec 7. PMID 21138487
- [Background] Wang Q, Lv H, Lu L, Ren P, Li L. Neonatal hypoxic-ischemic encephalopathy: emerging therapeutic strategies based on pathophysiologic phases of the injury. J Matern Fetal Neonatal Med. 2019 Nov;32(21):3685-3692. doi: 10.1080/14767058.2018.1468881. Epub 2018 May 2. PMID 29681183
- [Background] Hassell KJ, Ezzati M, Alonso-Alconada D, Hausenloy DJ, Robertson NJ. New horizons for newborn brain protection: enhancing endogenous neuroprotection. Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F541-52. doi: 10.1136/archdischild-2014-306284. Epub 2015 Jun 10. PMID 26063194
- [Background] McAdams RM, Juul SE. Neonatal Encephalopathy: Update on Therapeutic Hypothermia and Other Novel Therapeutics. Clin Perinatol. 2016 Sep;43(3):485-500. doi: 10.1016/j.clp.2016.04.007. Epub 2016 Jun 22. PMID 27524449
- [Background] Parikh P, Juul SE. Neuroprotective Strategies in Neonatal Brain Injury. J Pediatr. 2018 Jan;192:22-32. doi: 10.1016/j.jpeds.2017.08.031. Epub 2017 Oct 12. No abstract available. PMID 29031859
- [Background] Martinello K, Hart AR, Yap S, Mitra S, Robertson NJ. Management and investigation of neonatal encephalopathy: 2017 update. Arch Dis Child Fetal Neonatal Ed. 2017 Jul;102(4):F346-F358. doi: 10.1136/archdischild-2015-309639. Epub 2017 Apr 6. PMID 28389438
- [Background] Massaro AN, Wu YW, Bammler TK, Comstock B, Mathur A, McKinstry RC, Chang T, Mayock DE, Mulkey SB, Van Meurs K, Juul S. Plasma Biomarkers of Brain Injury in Neonatal Hypoxic-Ischemic Encephalopathy. J Pediatr. 2018 Mar;194:67-75.e1. doi: 10.1016/j.jpeds.2017.10.060. PMID 29478510
- [Background] Prempunpong C, Chalak LF, Garfinkle J, Shah B, Kalra V, Rollins N, Boyle R, Nguyen KA, Mir I, Pappas A, Montaldo P, Thayyil S, Sanchez PJ, Shankaran S, Laptook AR, Sant'Anna G. Prospective research on infants with mild encephalopathy: the PRIME study. J Perinatol. 2018 Jan;38(1):80-85. doi: 10.1038/jp.2017.164. Epub 2017 Nov 2. PMID 29095433
- [Derived] Tarocco A, Morciano G, Perrone M, Cafolla C, Ferre C, Vacca T, Pistocchi G, Meneghin F, Cocchi I, Lista G, Cetin I, Greco P, Garani G, Stella M, Natile M, Ancora G, Savarese I, Campi F, Bersani I, Dotta A, Tiberi E, Vento G, Chiodin E, Staffler A, Maranella E, Di Fabio S, Wieckowski MR, Giorgi C, Pinton P. Increase of Parkin and ATG5 plasmatic levels following perinatal hypoxic-ischemic encephalopathy. Sci Rep. 2022 May 12;12(1):7795. doi: 10.1038/s41598-022-11870-w. PMID 35551488